CLINICAL TRIAL: NCT00167089
Title: Effects of Early Treadmill Training on Ambulatory Ability in Stroke Patients: Electromyographic and Kinematic Analyses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: College of Medicine, National Taiwan University, College of Medicine, National Taiwan University
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 47s1
Record Dates: First submitted 2005-09-12; First posted 2005-09-14 (Estimated); Last update posted 2009-10-06 (Estimated); Status verified 2009-09

CONDITIONS: Stroke
Keywords: Stroke; Hemiplegia; Gait; Ambulation training; Neurologic physical therapy
MeSH Terms: conditions — Stroke; Hemiplegia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: Treadmill Training — Partian body weight support treadmill training, 30 min/day * 3 days /week

SUMMARY:
The purpose of this study is to explore an alternative approach that emphasizes task specificity and treadmill training for ambulation training of these patients.

DETAILED DESCRIPTION:
Restoration of independent ambulatory ability is one of the most common functional goals of patients with hemiplegia after stroke. Ambulation training, therefore, is an important part of physical therapy intervention for these patients. Conventional neurologic physical therapy for ambulation training, based sorely on neurophysiology, prohibits early ambulation experience after stroke in attempt to avoid the development of abnormal gait patterns. Such an approach has been shown to be limited in helping these patients regain independent ambulatory ability.

ELIGIBILITY:
Inclusion Criteria:

* between 40 and 75 years old
* first stroke with R't side hemiplegia due to middle cerebral artery occlusion and received acute treatment at NTUH
* being willing to sign an informed consent approved by the Human Subjects Committee of the National Taiwan University Hospital
* able to ambulate independently in parallel bars and having no independent ambulation ability outside parallel bars

Excursion criteria:

* having unstable vital sign, unconsciousness, or obvious cognitive, perception, and language impairment, and couldn't communicate with the experimenters
* having other neurological diseases, or moderate to severe neuromuscular or musculoskeletal or cardiovascular disorders, or disorders from systematic diseases other than stroke

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 1998-08; Primary Completion 2000-08 (Actual); Study Completion 2000-08 (Actual)

PRIMARY OUTCOMES:
To investigate walking speed and stride length as the representation of ambulation ability | 3 months

SECONDARY OUTCOMES:
To investigate the the co-activation duration between the activity of hamstring and quadriceps, and tibialis anterior and gastrocnemius joints, the level of symmetry in step length and stance/swing duration ratio between the affected and unaffected legs | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Pei-Fang Tang, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- School and Graduate Institute of Physical Therapy College of Medicine, National Taiwan University, Taipei, Province of China, Taiwan